CLINICAL TRIAL: NCT01980979
Title: Efficacy of Remodulin in Adults With Congenital Heart Disease (ACHD) and Pulmonary Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: University of California, Los Angeles (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, Jamil Aboulhosn, Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Remodulin in ACHD; IRB#12-001968 (Other: IRB#12-001968)
Record Dates: First submitted 2013-09-24; First posted 2013-11-11 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease,pulmonary hypertension,prostacyclin
MeSH Terms: conditions — Heart Defects, Congenital | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remodulin (Experimental): Subcutaneous (SQ) remodulin will be initiated at 1.25 ng/kg/min, and increased by 2-6 ng/kg/min weekly to a target dose of 40 ng/kg/min. If the initial infusion rate cannot be tolerated it will be reduced to 0.625 ng/kg/min. If subjects cannot tolerate the SQ therapy, we will attempt to switch to IV therapy.
  Interventions: Drug: Remodulin

INTERVENTIONS:
Drug: Remodulin — Subcutaneous (SQ) remodulin will be initiated at 1.25 ng/kg/min, and increased by 2-6 ng/kg/min weekly to a target dose of 40 ng/kg/min. If the initial infusion rate cannot be tolerated it will be reduced to 0.625 ng/kg/min. If subjects cannot tolerate the SQ therapy, we will attempt to switch to IV therapy.
  Other Names: treprostinil, tyvaso

SUMMARY:
The purpose of this study is to evaluate the efficacy of Remodulin in the treatment of adult patients with congenital heart disease and pulmonary hypertension. Baseline and post-treatment cardiopulmonary exercise tests will be performed.

DETAILED DESCRIPTION:
A prospective, open-label, non-randomized multi-center study is proposed to assess the efficacy of Remodulin in adults with congenital heart disease and pulmonary hypertension. Subjects will be enrolled at UCLA and Ohio State University (PI: Curt Daniels, MD). The study will involve a six month trial of continuous subcutaneous Remodulin therapy, with assessments conducted prior to initiation of therapy and at 1 and 6 months following initiation of therapy. A separate initiation visit will be scheduled after the baseline visit in order to provide subjects with comprehensive training in the use and care of the Remodulin drug delivery system.

Baseline and post-treatment (6 month) assessments will include a history and physical examination, cardiopulmonary exercise test, six minute walking distance, serum brain natriuretic peptide (BNP), a Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) quality of life survey, and subjective assessment of functional capacity (New York Heart Association (NYHA) scale). The interim (1 month) follow-up visit will include a thorough review of adverse events associated with Remodulin therapy, functional class assessment, six minute walk distance, and serum BNP.

Remodulin will be initiated at 1.25 ng/kg/min and increased by 2-6 ng/kg/min weekly to a target dose of 40 ng/kg/min. If the initial infusion rate cannot be tolerated it will be reduced to 0.625 ng/kg/min. Changes in drug dose will be at the discretion of the investigators following review of interim events. If necessary, the dose may be decreased by 2 ng/kg/min every two days as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Congenital heart disease with Pulmonary Arterial (PA) hypertension (repaired or unrepaired) defined as a mean resting directly measured Pulmonary Artery Pressure (PAP) of ≥35 mm Hg and/or doppler echo estimated PA systolic pressure ≥ 60 mm Hg.
* Patients already on phosphodiesterase type 5 inhibitor (PDE-5), Endothelin Receptor Antagonist (ERA), or inhaled prostacyclin are not excluded

Exclusion Criteria:

* Age < 18 years
* Current intravenous or subcutaneous prostacyclin therapy
* Resting systemic hypotension (Systolic blood pressure < 80 mm Hg)
* Women who are pregnant or may become pregnant (unwilling to utilize effective contraception), as well as nursing mothers
* Inability to ambulate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improved cardiopulmonary exercise test | 6 months
  Change in 6 minute walk distance after 6 months of escalating Subcutaneous (SQ) remodulin as compared to baseline.

SECONDARY OUTCOMES:
Improved overall cardiopulmonary variables | 1-6 months
  * Change in exercise duration (modified Bruce protocol)
  * Change in maximal oxygen consumption (VO2 max)
  * Change in minute ventilation- carbon dioxide production (VE/VCO2) ratio
  * Change in serum Brain Natriuretic Peptide (BNP) level
  * Change in quality of life as assessed by the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) survey
  * Change in resting oxygen saturation
  * Tricuspid Annular Plane Systolic Excursion (TAPSE)
  * Heart rate recovery

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Aboulhosn, MD, Principal Investigator — UCLA Health System
Locations (2):
- United States (2):
  - UCLA Medical Center, Los Angeles, California
  - Ohio State University/Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Background] Gomberg-Maitland M, Tapson VF, Benza RL, McLaughlin VV, Krichman A, Widlitz AC, Barst RJ. Transition from intravenous epoprostenol to intravenous treprostinil in pulmonary hypertension. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1586-9. doi: 10.1164/rccm.200505-766OC. Epub 2005 Sep 8. PMID 16151039
- [Background] Barst RJ, Galie N, Naeije R, Simonneau G, Jeffs R, Arneson C, Rubin LJ. Long-term outcome in pulmonary arterial hypertension patients treated with subcutaneous treprostinil. Eur Respir J. 2006 Dec;28(6):1195-203. doi: 10.1183/09031936.06.00044406. Epub 2006 Aug 9. PMID 16899485
- [Background] Tapson VF, Gomberg-Maitland M, McLaughlin VV, Benza RL, Widlitz AC, Krichman A, Barst RJ. Safety and efficacy of IV treprostinil for pulmonary arterial hypertension: a prospective, multicenter, open-label, 12-week trial. Chest. 2006 Mar;129(3):683-8. doi: 10.1378/chest.129.3.683. PMID 16537868
- [Background] Simonneau G, Barst RJ, Galie N, Naeije R, Rich S, Bourge RC, Keogh A, Oudiz R, Frost A, Blackburn SD, Crow JW, Rubin LJ; Treprostinil Study Group. Continuous subcutaneous infusion of treprostinil, a prostacyclin analogue, in patients with pulmonary arterial hypertension: a double-blind, randomized, placebo-controlled trial. Am J Respir Crit Care Med. 2002 Mar 15;165(6):800-4. doi: 10.1164/ajrccm.165.6.2106079. PMID 11897647
- See also: UCLA Adult Congenital Heart Disease Center — http://heart.ucla.edu/achdc